CLINICAL TRIAL: NCT04235049
Title: Elimination of HCV Through Linkage and In Prison Treatment of Incarcerated Populations
Brief Title: Elimination of HCV Through Linkage and In Prison Treatment of Incarcerated Populations (ECLIPSE)
Acronym: ECLIPSE
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Department of Corrections unable to support study at this time and find agreement on publication issue.
Sponsor: University of Maryland, Baltimore (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); Maryland Department of Public Safety and Correctional Services (Unknown)
Responsible Party: Principal Investigator, Elana Rosenthal, Assistant Professor, University of Maryland, Baltimore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HP-00088498
Record Dates: First submitted 2020-01-10; First posted 2020-01-21 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-04

CONDITIONS: HCV Infection
Keywords: HCV infection; Incarcerated individuals
MeSH Terms: conditions — Hepatitis C | interventions — glecaprevir and pibrentasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- In prison treatment arm (No Intervention): Of patients who achieved SVR, 100 inmates will be enrolled for long-term monitoring for re-infection after they have completed treatment. Patients will be seen every 6 months to test for reinfection, however they will not be subject to any medical or behavioral interventions through the study team. Limited opioid agonist therapy may be available as per the standard practice of the DOC, however syringe exchange and other harm reduction services will not be accessible to inmates, per DOC policy.
- Community Linkage - Rapid Initiation Arm (Active Comparator): The rapid initiation group will receive HCV medication immediately upon release from prison/jail.
  Interventions: Drug: Glecaprevir/pibrentasvir
- Community Linkage - Clinic-Based Initiation Arm (Active Comparator): The group will receive medication after attending first ANCHOR clinic visit.
  Interventions: Drug: Glecaprevir/pibrentasvir
- In prison - Retrospective Review (No Intervention): a retrospective review of de-identified available data provided by the DOC for all patients previously treated with DAAs through standard of care in the DOC will be reviewed for rates of SVR.

INTERVENTIONS:
Drug: Glecaprevir/pibrentasvir — Treatment for HCV Infection
  Arms: Community Linkage - Clinic-Based Initiation Arm; Community Linkage - Rapid Initiation Arm

SUMMARY:
Hepatitis C (HCV) is a chronic infection with significant morbidity and mortality. The development of directly acting antivirals (DAA) has dramatically improved the cure rate of HCV treatment. People who experience incarceration are disproportionately infected and often involved in ongoing transmission of disease. However, despite availability of effective treatment, people who experience incarceration are often unable to access this curative therapy, and are often not readily engaged in medical care upon release. This perpetuates transmission and progression of disease in an incredibly high risk, marginalized population. Therefore, in order to effectively eliminate HCV, it is imperative that the epidemic of HCV in prisons is addressed, and that models of care are established for treatment of HCV in incarcerated individuals, both during and after incarceration.

As such, the investigators propose a comprehensive model of care to engage incarcerated individuals in treatment of HCV upon release from prison. This care is provided in conjunction with collocated services to prevent HCV reinfection, including opioid agonist therapy. This pilot trial will demonstrate whether a comprehensive model of care can effectively cure HCV in recently incarcerated individuals, while simultaneously treating opioid use disorder and preventing HCV reinfection.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 18 years old
2. Able and willing to sign informed consent
3. For the community linkage arm: Chronically infected with HCV, defined as any individual with documentation of positive HCV antibody and positive HCV RNA test (HCV RNA of 2,000 IU/mL or greater).
4. For the community linkage arm: ineligible for treatment through the prison/jail without a known sentence longer than 9 months, as of consent date
5. For the in-prison arm: Achievement of SVR through the previous standard of care treatment through the DOC

Exclusion Criteria:

1. Decompensated cirrhosis (Child-Pugh B or C)
2. Pregnant or breastfeeding women
3. For community linkage arm: Prior treatment with a direct acting antiviral regimen
4. For community linkage arm: Any co-medications that are contraindicated or not recommended for concomitant use with glecaprevir-pibrentasvir
5. Poor venous access not allowing screening laboratory collection
6. Have any condition that the investigator considers a contraindication to study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2022-03-30 (Estimated); Study Completion 2024-10-30 (Estimated)

PRIMARY OUTCOMES:
Sustained Virologic Response (SVR) in the community linkage arm | 6 months after treatment
  Absence of plasma HCV RNA levels 70 days or greater after completing direct acting antiviral therapy.

SECONDARY OUTCOMES:
Retrospective rates of SVR in the In prison arm | 6 months after treatment
  Absence of plasma HCV RNA levels 70 days or greater after completing direct acting antiviral therapy.
Treatment Initiation Rates | 6 months
  Rates of treatment initiation in the CL arm (defined as taking one dose of direct acting antiviral)
OAT uptake Rates | 12 months
  Rates of OAT uptake in the CL arm (defined as completion of OAT induction)
HCV Reinfection Rates | 24 months
  Reinfection (defined as documentation of infection with a different HCV genotype than at baseline before treatment, or if the same genotype, viremia after SVR determination, or phylogenetic analysis shows a different virus strain than the pre treatment baseline strain)
Comparison between Rapid Initiation and Clinic-base Initiation | 24 months
  Comparative efficacy of rapid initiation (RI) and clinic-based initiation (CB) arms, comparing the rates of SVR in patients who were randomized to the RI arm compared to patients randomized to the CB arm.

CONTACTS AND LOCATIONS:
Overall Officials: Elana Rosenthal, MD, Principal Investigator — University of Maryland, Baltimore
Locations (1):
- Baltimore City Detention Center, Baltimore, Maryland, United States